CLINICAL TRIAL: NCT05748093
Title: Improving Osimertinib Exposure and Cost-effectiveness Using Pharmacokinetic Boosting With Cobicistat (OSIBOOST 2)
Brief Title: Improving Osimertinib Exposure and Cost-effectiveness Using Pharmacokinetic Boosting With Cobicistat
Acronym: OSIBOOST 2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSIBOOST 2; 2023-505700-35-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-02; First posted 2023-02-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Osimertinib; Cobicistat; Pharmacokinetics; Boosting; Non-small Cell Lung Cancer; CNS metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cobicistat

STUDY DESIGN:
Intervention Model Description: This study will involve two cohorts, which will both receive PK-boosting, but for different purposes, and with different primary outcomes. The cohorts will not be compared, and there will be no cross-over between cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Adjusting osimertinib treatment plans with concomitant pk-boosting (Experimental): Feasibility of using pharmacokinetic boosting and TDM to individualize treatment plans and dosage for osimertinib, in patients with advanced NSCLC with mutated EGFR. In this cohort, patients will receive cobicistat for pharmacokinetic boosting of standard osimertinib treatment. Afterwards, they will receive personalised treatment plans, guided by therapeutic drug monitoring.
  Interventions: Drug: Cobicistat
- Cohort 2: Improving osimertinib CNS penetration in patients with neurometastases (Experimental): Assessing whether pharmacokinetic boosting can improve CNS penetration of osimertinib, in patients with advanced NSCLC with mutated EGFR with asymptomatic CNS oligoprogression. Patients who experience progressive disease intracranially, are sometimes dose-escalated to try and improve osimertinib intracranial exposure. This study will look to demonstrate the feasibility of using a PK-booster instead, potentially providing patients the benefits of higher intracranial treatment efficacy, without needing to take extra osimertinib.
  Interventions: Drug: Cobicistat

INTERVENTIONS:
Drug: Cobicistat — Feasibility of pharmacokinetic boosting using cobicistat for personalized treatment strategies for osimertinib.
  Other Names: Tybost

SUMMARY:
The goal of this clinical trial is to assess the feasibility of pharmacokinetically boosting osimertinib using cobicistat in order to improve osimertinib exposure in individual patients with advanced NSCLC (Non-Small Cell Lung Cancer) with mutated EGFR (Epidermal Growth Factor Receptor). The main questions it aims to answer are:

* Cohort 1: Does concurrent use of osimertinib and cobicistat allow for osimertinib weekly intake reductions? If so, how much can the intake be reduced while retaining clinically effective exposure?
* Cohort 2: Does concurrent use of osimertinib and cobicistat allow for improved penetration of osimertinib in the central nervous system, in patients with CNS (central nervous system) oligoprogression?

Participants who are taking osimertinib in regular care will receive cobicistat in addition to their other medication. They will undergo blood sampling to measure the amount of osimertinib in blood, and measure the effect of boosting. Additionally, in cohort 1 patients will be dose-reduced if their exposure levels allow.

DETAILED DESCRIPTION:
In 2016 Osimertinib was registered for the treatment of patients with metastatic Non-Small Cell Lung Cancer (NSCLC) with an activating Epidermal Growth Factor Receptor (EGFR) mutation, initially only for patients with the T790M resistance mutation, but since 2018 also in the first line treatment. Use of osimertinib in the first line provides improved overall survival and progression-free survival, more potent efficacy against brain metastases, and better tolerability compared to older generation EGFR tyrosine kinase inhibitors (EGFR-TKIs). The downside of osimertinib is that -like many new anticancer agents- it is highly expensive (over €70 000 per patient per year in the Netherlands). In a period of five years, healthcare costs associated with expensive medication have risen from €1.71 billion to €2.46 billion per year in the Netherlands. The Dutch Cancer Society has warned that this astronomical cost increase will start to suffocate the national health care budget. In order to safeguard sustained affordability and accessibility of oncological healthcare, improving cost-effectiveness of available drugs is of paramount importance. In a previous study, we have demonstrated that osimertinib exposure may be boosted, through concomitant use of cobicistat, as a result of CYP3A4 inhibition. We now aim to apply pharmacokinetic (PK) boosting in order to improve osimertinib exposure and cost-effectiveness, without impacting treatment efficacy and safety.

This trial is designed to study whether pharmacokinetic boosting may alleviate these issues. In the first cohort, we will assess whether PK-boosting is able to reduce the amount of osimertinib which a patient needs to take. In order to assess this, the patient will receive cobicistat (the booster drug) and we will measure the amount of osimertinib and its metabolite in blood. Afterwards, the researchers and physicians may calculate how much osimertinib a patient actually needs. Ideally this will both reduce the amount of osimertinib that a patient needs to take, as well as reduce the price-tag of the overall treatment. In the second cohort, we will assess whether PK-boosting is a viable alternative to dose-doubling osimertinib. Some patients with NSCLC develop progressive CNS metastases despite osimertinib therapy. There is an indication that increasing the osimertinib dosage to double the standard therapy might provide longer/better treatment efficacy in these patients. Because of the tremendous cost associated with double-dosing osimertinib, most health care insurance providers in the Netherlands do not cover this therapy. In cohort 2 we look to find out whether PK-boosting might provide a similar effect to increasing the dosage, for a far more affordable price-tag.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this cohort 1, a subject must meet all of the following criteria:

* The patient is set to receive osimertinib 80 mg QD as part of their standard treatment plan
* The patient has a World Health Organization (WHO) Performance Status (PS) of ≤2.
* The patient is 18 years or older
* The patient is able and willing to sign informed consent
* The patient is able and willing to undergo blood sampling
* The patient has non-squamous advanced EGFR-mutated NSCLC with no signs of imminent progression (CT confirmed). If the patient does have signs of progression, they are only eligible if their treating physician deems the treatment to be appropriate beyond progression.
* The patient consents to their blood being analysed for CYP3A-genotype

In order to be eligible to participate in this cohort 2, a subject must meet all of the following criteria:

* The patient is set to receive osimertinib 80 mg QD as part of their standard treatment plan
* The patient has a World Health Organization (WHO) Performance Status (PS) of ≤2.
* The patient is 18 years or older
* The patient is able and willing to sign informed consent
* The patient is able and willing to undergo blood sampling
* The patient has non-squamous EGFR-mutated NSCLC with radiologically confirmed progressive (RECIST v1.1), but asymptomatic intracranial metastasis, not in an eloquent area (to be discussed with neurologist). Furthermore, the disease is controlled extracranially (no RECIST v1.1 progression).

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study:

* The patient does not take any other drug which is known to strongly inhibit CYP3A4/CYP3A5 activity
* The patient does not take any other drug which is metabolized by CYP3A4/CYP3A5 and which has a small therapeutic window
* The patient does not take any drug or product which may otherwise affect CYP3A4/CYP3A5 metabolic activity
* The patient does not have impaired gastrointestinal function
* The patient is neither pregnant nor breastfeeding
* The patient does not have any contra-indication for cobicistat prescription, as listed in the summary of product characteristics for cobicistat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 primary end-point: Dose modification feasibility | 2-18 months after intervention initiation
  This cohort aims to demonstrate feasibility and clinical applicability of PK-boosting in the oncological setting. PK-boosting will increase osimertinib availability in plasma. When the availability is increased, a patient will require less osimertinib to achieve the same effect. Therefore, they can be dose-reduced in order to restore them to their normal exposure. In order for this treatment to be considered feasible, the following conditions need to be met: a patient needs to have a stable osimertinib exposure when using the PK-booster, and the patient needs to be dose-modified as a result. The primary endpoint will describe the amount of patients who have: stable exposure; similar to their respective baseline; while using concomitant pk-boosting therapy and a dose modified osimertinib treatment plan; without experiencing significant toxicity. The aim is for this treatment strategy to be considered feasible for at least 75% of patients.
Cohort 2 primary end-point: Disease Control Rate at 12 weeks | 12 weeks after intervention initiation
  This cohort aims to provide improved treatment efficacy in patients with intracranial metastases from NSCLC. Osimertinib penetration in the CNS is much better than that of older generation TKIs, but it is still only 1,49%. Many patients with NSCLC end up developing CNS metastases, a condition known for its dismal prognosis. Currently the only way to increase osimertinib CNS penetration is through dose-escalation: a strategy which causes a tremendous increase in treatment-related toxicity. This cohort looks to improve CNS penetration of osimertinib through the use of a PK-booster (cobicistat). In order to assess treatment efficacy, a MRI will be taken at the start of the trial, and after 12 weeks. A neuro-radiology panel will then assess metastatic response rate. This metastatic response rate will be compared to historical data in order to assess the intracranial treatment efficacy.

SECONDARY OUTCOMES:
Cohort 1 secondary end-point: plasma concentrations of osimertinib and AZ5104 | 2-18 months after intervention initiation
  In order to assess the extent of pharmacokinetic boosting in plasma, the plasma concentrations of osimertinib and AZ5104 (metabolite) will be determined.
Cohort 1 secondary end-point: safety set | 2-18 months after intervention initiation
  Number of (serious) adverse events as graded by CTCAE
Cohort 1 secondary end-point: Cost-effectiveness analysis | 2-18 months after intervention initiation
  If in cohort 1 the overall treatment is considered "feasible". An assessment of overall average treatment cost per patient per day will be made for the experimental treatment plan. This will be compared to the current standard treatment cost using a Health-Technology Assessment (HTA). If efficacy endpoints cannot be determined, but the trial treatment is considered "feasible", then the trial treatment will be assessed as "non-inferior" (as the TDM-strategy looks to maintain similar drug exposure).
Cohort 1 secondary end-point: CYP3A predictiveness for osimertinib exposure | 2-18 months after intervention initiation
  Assessing predictiveness of CYP3A-polymorphism for osimertinib exposure. This will be done by statistically comparing osimertinib exposure for patient groups with different genotypes.
Cohort 2 secondary end-point: plasma concentrations of osimertinib and AZ5104 | 12 weeks after intervention initiation
  In order to assess the extent of pharmacokinetic boosting in plasma, the plasma concentrations of osimertinib and AZ5104 (metabolite) will be determined.
Cohort 2 secondary end-point: safety set | 12 weeks after intervention initiation
  Number of (serious) adverse events as graded by CTCAE

OTHER OUTCOMES:
Cohort 1 exploratory end-point: Comparison of progression-free survival to historical data | 2-18 months after intervention initiation
  The efficacy of palliative cancer treatment is mostly assessed through progression-free survival. Because of its explorative nature, this trial will not be equipped to provide a statistical analysis of both treatments. Therefore average progression-free survival will be compared numerically to historical data, in order to provide an indication of treatment efficacy.
Cohort 2 exploratory end-point: Comparison of Progression-free Survival to historical data | 12 weeks after intervention initiation
  The efficacy of palliative cancer treatment is mostly assessed through progression-free survival. Because of its explorative nature, this trial will not be equipped to provide a statistical analysis of both treatments. Therefore average progression-free survival will be compared numerically to historical data, in order to provide an indication of treatment efficacy.
Cohort 2 exploratory end-point: Extracranial disease control | 12 weeks after intervention initiation
  Disease control rate for extracranial disease, as assessed by thoracic imaging
Cohort 2 exploratory end-point: Osimertinib and AZ5104 concentrations in cerebrospinal fluid. | 12 weeks after intervention initiation
  On a voluntary basis, patients may opt to undergo lumbar punctures, to allow for determination of osimertinib and AZ5104 (metabolite) exposure in the brain liquor (cerebrospinal fluid). This will be a purely descriptive analysis. This technique might help to shed light on how well osimertinib and its metabolite is able to reach CNS metastases. Because of the invasive nature of the analysis, lumbar punctures will be considered optional, and not required for trial participation.
Cohort 2 exploratory end-point: Liquid biopsy measurements of resistance mutations in cerebrospinal fluid | 12 weeks after intervention initiation
  On a voluntary basis, patients may opt to undergo lumbar punctures, to allow for determination of tumor-cell genotype and the presence of resistance mutations through liquid biopsy analysis. This will be a purely descriptive analysis. This technique might help to shed light on how resistance develops in CNS metastases. Because of the invasive nature of the analysis, lumbar punctures will be considered optional, and not required for trial participation.

CONTACTS AND LOCATIONS:
Overall Officials: Lizza Hendriks, MD, PhD, Principal Investigator — Maastricht University Medical Centre+
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Veelen A, Gulikers J, Hendriks LEL, Dursun S, Ippel J, Smit EF, Dingemans AC, van Geel R, Croes S. Pharmacokinetic boosting of osimertinib with cobicistat in patients with non-small cell lung cancer: The OSIBOOST trial. Lung Cancer. 2022 Sep;171:97-102. doi: 10.1016/j.lungcan.2022.07.012. Epub 2022 Jul 25. PMID 35933915
- [Background] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359